CLINICAL TRIAL: NCT04525950
Title: Robotized Computer Navigation Versus Conventional Technique in Total Knee Replacement. A Randomized, Clinical and Radiostereometric Trial.
Brief Title: Robotized Navigation Compared to Conventional Technique in Total Knee Replacement
Acronym: NavioRCT
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Haukeland University Hospital (Other)
Collaborators: University of Bergen (Other); Haugesund Rheumatism Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2020/68448
Record Dates: First submitted 2020-08-17; First posted 2020-08-25 (Actual); Last update posted 2025-03-14 (Actual); Status verified 2024-10

CONDITIONS: Arthritis, Degenerative; Osteo Arthritis Knee
MeSH Terms: conditions — Osteoarthritis | interventions — Congresses as Topic

STUDY DESIGN:
Intervention Model Description: Randomized, blinded (patient and outcomes assessor), clinical and radiostereometric trial
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Participants are blinded as the Navio system will be switched on at all operations, the outcomes assessors, statisticians and co-researchers will not get access to the randomization information.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Navio (Experimental): Using the new technology during surgery
  Interventions: Procedure: Navio
- Conventional (Active Comparator): Using the conventional surgical instruments
  Interventions: Procedure: Conventional

INTERVENTIONS:
Procedure: Navio — New generation computer navigation with haptics and robotics
  Arms: Navio
Procedure: Conventional — Total knee arthroplasty using conventional instruments
  Arms: Conventional

SUMMARY:
Navio is a new generation of computer navigation systems allowing intraoperative navigation of the bone cuts relative to both ligaments and skeletal axes, prior to bone removal. An improved accuracy is incorporated by the use of robotics in a burr for bone removal.

This study investigates whether this advanced technology leads to better clinical or radiostereometric results, by comparing one group operated with Navio to another group operated with conventional technique.

DETAILED DESCRIPTION:
Background:

The scientific foundation of total knee replacement (TKR) surgery is incomplete. As a national governor of joint replacements, the Norwegian Arthroplasty Register is obligated to strict regulations, demanding high levels of evidence for implants and instruments utilized by Norwegian surgeons. It is well known that 15-20% of patients with a TKR, are dissatisfied. Nevertheless, only a small proportion of these patients have revision surgery.

In this randomized, clinical trial we will use the Journey II BCS total knee system, with a more native anatomical design, intended to improve the kinematics and functional outcomes by mimicking a native knee, with respect to geometry and its interplay with the ligaments and soft tissue envelope of the knee (i.e. the biomechanics; stability, joint line, off-set, sizing etc.). To achieve an optimal placement of the implant, the surgeon needs to assess a lot of information (experience) during the surgical procedure. To secure this process, and to make sure all aspects are taken into account, with respect to an optimal positioning and ligament balancing, the computer navigation technique may offer valuable input, with further enhancement of the accuracy and precision using precision tools like the Navio from Smith & Nephew. The Navio system combines robotics and computer navigation, and represents the newest technology within surgical robotics and haptics. This trial is important in the mandatory evaluation process needed, before introducing new technology into orthopaedic surgery, on a larger scale.

Methods:

The surgeons involved have been trained at a wet lab, and on saw bones, before utilizing this tool in a live setting. After the introduction period, the training will continue in a clinical setting until the surgeons have operated at least 20 Navio assisted cases each, followed by a pilot study of 10 patients. All patients will be randomized to either Navio or Conventional technique.

Surgical method: A tourniquet is used. All implant components are cemented (Palacos R+G bone cement is utilized 10 minutes after retrieval from a 4 degrees Celsius refrigerator). Standard para-patellar approach. ACL and PCL are removed. Closing of the wound and capsule in mid-flexion position, Quill for the capsule, Vicryl for the subcutaneous tissue, continuous overlapping mattress with Ethilon suture for the skin. No drainage. Wrapping of the entire limb with elastic dressings for the first 48 hours. Prophylactic antibiotics and anticoagulants are given. Tranexamic acid to reduce bleeding. Postop pain medication: gabapentin, acetaminophen, naproxen, femoral triangle nerve block (repeated next day if needed).

For the conventional group: The rotational alignment is set according to Whiteside's line, and intramedullary rods with 5, 6 or 7 degrees valgus, are selected for the distal femoral cut (dependent on pre-operatively measured angles on long radiographs (hip-knee-ankle). The entry hole of the rod is plugged with bone from the femur to reduce bleeding from the intramedullary canal. The tibial component (metal) is positioned with a 3 degrees posterior slope.

For the Navio group: The cuts are navigated to optimize ligament balance in flexion and extension, and adjusted for mid-flexion instability when needed. A difference of less than 4 mm between lateral and medial gaps is accepted when the laxity is on the lateral side, preferably in flexion. However, if the gap balancing technique suggests a deviation from mechanical alignment of more than 2 degrees of valgus or 4 degrees of varus, the suggestion is overruled by the mechanical alignment (maximum 2 degrees valgus, less than 4 degrees varus).

Sample size calculations: To detect a clinically important difference of 0.17 in the rate of "high responders" and "non-responders" (OMERACT-OARSI criteria) to the Navio, with a standard deviation of 20, power 80% and a 0.05 significance level, a total of 194 patients must be included in the trial (97 patients in each group). The calculations are based on data from a previous study, by Petursson et al, JBJS Am 2018. When 10% eventual drop-outs are taken into account, the total number of patients to be included is 214 (107 patients in each group).

A large number of patients is important, as the expected difference between the groups is small. A small difference may be less clinically relevant, however, may contribute to an overall better outcome for the patients in total. A small improvement of the tools combined with other small improvements may add up to be clinically important in the end. Small trials with no significant differences may disqualify important small improvements, thus stopping any further development in the field. Consequently, large clinical trials will be valuable.

A radiostereometric analysis constitutes a separate study of the trial. A clinically relevant difference of 0.1 mm between the groups will be detected with a standard deviation of 0.1, power 80% and significance level 0.05, if 17 patients are included in each group. Including eventual drop-outs and an expectation of some failures due to the technically challenging investigation method (the RSA), a total of 30 patients will be included in each group. RSA radiographs will be collected within the first week after the operation, at 3 months, 1 year, 2 years and 5 years follow-ups.

The trial is approved by the regional ethics committee and the data inspectorate of Norway.

ELIGIBILITY:
Inclusion Criteria:

* Degenerative knee in need of a total knee arthroplasty
* Recruited from the hospital's waiting list
* Informed consent

Exclusion Criteria:

* Severe systemic illness
* Infections
* Severe neurological dysfunction
* Severe cancer disease
* Severe incompensated heart failure
* Severe incompensated lung disease
* Dementia
* Previous fracture or deformity of the limb, making the use of an intramedullary rod impossible (same side hip or ankle implant is not to be excluded if the rod unaffectedly reaches more than the first half of the femoral canal)

Ages: 45 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 214 (Estimated)
Dates: Start 2020-09-07 (Actual); Primary Completion 2023-05-01 (Actual); Study Completion 2031-12-31 (Estimated)

PRIMARY OUTCOMES:
Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) high responders | 3 months
  Difference in rate (0.00-1.00) of high responders (calculated from KOOS)
WOMAC high responders | 1 year
  Difference in rate (0.00-1.00) of high responders (calculated from KOOS)
WOMAC high responders | 2 years
  Difference in rate (0.00-1.00) of high responders (calculated from KOOS)
WOMAC high responders | 5 years
  Difference in rate (0.00-1.00) of high responders (calculated from KOOS)
Radiostereometric migration | 1 year
  Maximum total point of motion MTPM (millimeters), (includes only first 60 patients)
Radiostereometric migration | 2 years
  Maximum total point of motion MTPM (millimeters), (includes only first 60 patients)
Radiostereometric migration | 5 years
  Maximum total point of motion MTPM (millimeters), (includes only first 60 patients)

SECONDARY OUTCOMES:
Knee injury and osteoarthritis outcome score (KOOS) | 3 months
  Symptoms, Stiffness, Pain, Activity of daily living, Sports, Quality of life subscores (0(worse)-100(better))
Knee injury and osteoarthritis outcome score (KOOS) | 1 year
  Symptoms, Stiffness, Pain, Activity of daily living, Sports, Quality of life subscores (0-100)
Knee injury and osteoarthritis outcome score (KOOS) | 2 years
  Symptoms, Stiffness, Pain, Activity of daily living, Sports, Quality of life subscores (0-100)
Knee injury and osteoarthritis outcome score (KOOS) | 5 years
  Symptoms, Stiffness, Pain, Activity of daily living, Sports, Quality of life subscores (0-100)
Knee society score (KSS) | 3 months
  Knee society score, knee score (0(worse)-100(better)) and function score (0(worse)-100(better))
Knee society score (KSS) | 1 year
  Knee society score, knee score (0-100) and function score (0-100)
Knee society score (KSS) | 2 years
  Knee society score, knee score (0-100) and function score (0-100)
Knee society score (KSS) | 5 years
  Knee society score, knee score (0-100) and function score (0-100)
EQ-5D | 3 months
  Euroqol, quality of life (0(worse)-100(better))
EQ-5D | 1 year
  Euroqol, quality of life (0-100)
EQ-5D | 2 years
  Euroqol, quality of life (0-100)
EQ-5D | 5 years
  Euroqol, quality of life (0-100)
Visual analogue scale (VAS) | pre-op, 3 months, 1 year, 2 years, 5 years
  Visual Analogue Scale pain (0(worse)-100(better))
Forgotten Joint Score (FJS) | 3 months
  Forgotten Joint Score (0(worse)-100(better))
Forgotten Joint Score (FJS) | 1 year
  Forgotten Joint Score (0-100)
Forgotten Joint Score (FJS) | 2 years
  Forgotten Joint Score (0-100)
Forgotten Joint Score (FJS) | 5 years
  Forgotten Joint Score (0-100)
Maximum climb-up test | 3 months
  Height (cm) of one stair climbed with affected/operated limb (no pulling by hands)
Maximum climb-up test | 1 year
  Height (cm) of one stair climbed with affected/operated limb (no pulling by hands)
Anchor questions | 2 years
  Are you satisfied with the outcome? Would you do it again?
Anchor questions | 5 years
  Are you satisfied with the outcome? Would you do it again?
Timed 40 meters walking test | 3 months
  Time spent walking 40 meters
Timed 40 meters walking test | 1 year
  Time spent (in seconds) walking 40 meters
Chair test 30 seconds | 3 months
  number of repetitions from sitting to standing position during 30 seconds
Chair test 30 seconds | 1 year
  number of repetitions from sitting to standing position during 30 seconds

OTHER OUTCOMES:
Position of the implant on radiographs, coronal and sagittal plane | 3 months
  Femoral/tibial components: varus/valgus and flexion/extension, off-set of the femoral component

CONTACTS AND LOCATIONS:
Overall Officials: Ove Furnes, MD/PhD, Study Chair — University of Bergen
Locations (2):
- Norway (2):
  - Haugesund sanitetsforenings revmatismesykehus, Haugesund, Haugesund
  - Haukeland university hospital, Bergen

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Batailler C, White N, Ranaldi FM, Neyret P, Servien E, Lustig S. Improved implant position and lower revision rate with robotic-assisted unicompartmental knee arthroplasty. Knee Surg Sports Traumatol Arthrosc. 2019 Apr;27(4):1232-1240. doi: 10.1007/s00167-018-5081-5. Epub 2018 Jul 31. PMID 30066017
- [Background] Petursson G, Fenstad AM, Gothesen O, Dyrhovden GS, Hallan G, Rohrl SM, Aamodt A, Furnes O. Computer-Assisted Compared with Conventional Total Knee Replacement: A Multicenter Parallel-Group Randomized Controlled Trial. J Bone Joint Surg Am. 2018 Aug 1;100(15):1265-1274. doi: 10.2106/JBJS.17.01338. PMID 30063588
- [Background] Robinson PG, Clement ND, Hamilton D, Blyth MJG, Haddad FS, Patton JT. A systematic review of robotic-assisted unicompartmental knee arthroplasty: prosthesis design and type should be reported. Bone Joint J. 2019 Jul;101-B(7):838-847. doi: 10.1302/0301-620X.101B7.BJJ-2018-1317.R1. PMID 31256672
- [Background] Bollars P, Boeckxstaens A, Mievis J, Kalaai S, Schotanus MGM, Janssen D. Preliminary experience with an image-free handheld robot for total knee arthroplasty: 77 cases compared with a matched control group. Eur J Orthop Surg Traumatol. 2020 May;30(4):723-729. doi: 10.1007/s00590-020-02624-3. Epub 2020 Jan 16. PMID 31950265
- [Background] Roos EM, Roos HP, Lohmander LS, Ekdahl C, Beynnon BD. Knee Injury and Osteoarthritis Outcome Score (KOOS)--development of a self-administered outcome measure. J Orthop Sports Phys Ther. 1998 Aug;28(2):88-96. doi: 10.2519/jospt.1998.28.2.88. PMID 9699158
- [Background] Roos EM, Roos HP, Ekdahl C, Lohmander LS. Knee injury and Osteoarthritis Outcome Score (KOOS)--validation of a Swedish version. Scand J Med Sci Sports. 1998 Dec;8(6):439-48. doi: 10.1111/j.1600-0838.1998.tb00465.x. PMID 9863983
- [Background] Heijbel S, Naili JE, Hedin A, W-Dahl A, Nilsson KG, Hedstrom M. The Forgotten Joint Score-12 in Swedish patients undergoing knee arthroplasty: a validation study with the Knee Injury and Osteoarthritis Outcome Score (KOOS) as comparator. Acta Orthop. 2020 Feb;91(1):88-93. doi: 10.1080/17453674.2019.1689327. Epub 2019 Nov 12. PMID 31711349
- [Background] Ko V, Naylor JM, Harris IA, Crosbie J, Yeo AE. The six-minute walk test is an excellent predictor of functional ambulation after total knee arthroplasty. BMC Musculoskelet Disord. 2013 Apr 24;14:145. doi: 10.1186/1471-2474-14-145. PMID 23617377
- [Background] Unver B, Kalkan S, Yuksel E, Kahraman T, Karatosun V. Reliability of the 50-foot walk test and 30-sec chair stand test in total knee arthroplasty. Acta Ortop Bras. 2015 Jul-Aug;23(4):184-7. doi: 10.1590/1413-78522015230401018. PMID 26327798
- [Background] Nyberg LA, Hellenius ML, Wandell P, Kowalski J, Sundberg CJ. Maximal step-up height as a simple and relevant health indicator: a study of leg muscle strength and the associations to age, anthropometric variables, aerobic fitness and physical function. Br J Sports Med. 2013 Oct;47(15):992-7. doi: 10.1136/bjsports-2013-092577. Epub 2013 Aug 21. PMID 23966416
- [Background] Gothesen O, Espehaug B, Havelin LI, Petursson G, Hallan G, Strom E, Dyrhovden G, Furnes O. Functional outcome and alignment in computer-assisted and conventionally operated total knee replacements: a multicentre parallel-group randomised controlled trial. Bone Joint J. 2014 May;96-B(5):609-18. doi: 10.1302/0301-620X.96B5.32516. PMID 24788494
- [Background] Inui H, Taketomi S, Yamagami R, Shirakawa N, Kawaguchi K, Tanaka S. The Relationship between Soft-Tissue Balance and Intraoperative Kinematics of Guided Motion Total Knee Arthroplasty. J Knee Surg. 2019 Jan;32(1):91-96. doi: 10.1055/s-0038-1636545. Epub 2018 Mar 7. PMID 29514366
- [Background] Iriuchishima T, Ryu K. Bicruciate Substituting Total Knee Arthroplasty Improves Stair Climbing Ability When Compared with Cruciate-Retain or Posterior Stabilizing Total Knee Arthroplasty. Indian J Orthop. 2019 Sep-Oct;53(5):641-645. doi: 10.4103/ortho.IJOrtho_392_18. PMID 31488934
- [Background] Harris AI, Christen B, Malcorps JJ, O'Grady CP, Kopjar B, Sensiba PR, Vandenneucker H, Huang BK, Cates HE, Hur J, Marra DA. Midterm Performance of a Guided-Motion Bicruciate-Stabilized Total Knee System: Results From the International Study of Over 2000 Consecutive Primary Total Knee Arthroplasties. J Arthroplasty. 2019 Jul;34(7S):S201-S208. doi: 10.1016/j.arth.2019.02.011. Epub 2019 Feb 14. PMID 31031156
- [Background] Kono K, Inui H, Tomita T, Yamazaki T, Taketomi S, Sugamoto K, Tanaka S. Bicruciate-stabilised total knee arthroplasty provides good functional stability during high-flexion weight-bearing activities. Knee Surg Sports Traumatol Arthrosc. 2019 Jul;27(7):2096-2103. doi: 10.1007/s00167-019-05375-9. Epub 2019 Apr 10. PMID 30972466
- [Background] Di Benedetto P, Buttironi MM, Magnanelli S, Cainero V, Causero A. Comparison between standard technique and image-free robotic technique in medial unicompartmental knee arthroplasty. Preliminary data. Acta Biomed. 2019 Dec 5;90(12-S):104-108. doi: 10.23750/abm.v90i12-S.8994. PMID 31821293
- [Background] Unver B, Kahraman T, Kalkan S, Yuksel E, Karatosun V. Reliability of the six-minute walk test after total hip arthroplasty. Hip Int. 2013 Nov-Dec;23(6):541-5. doi: 10.5301/hipint.5000073. Epub 2013 Aug 6. PMID 23934905
- [Background] Petursson G, Fenstad AM, Gothesen O, Haugan K, Dyrhovden GS, Hallan G, Rohrl SM, Aamodt A, Nilsson KG, Furnes O. Similar migration in computer-assisted and conventional total knee arthroplasty. Acta Orthop. 2017 Apr;88(2):166-172. doi: 10.1080/17453674.2016.1267835. Epub 2016 Dec 20. PMID 27996349